CLINICAL TRIAL: NCT03832972
Title: Variation in Performance During Menstrual Cycle
Brief Title: Performance During Menstrual Cycle
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Team Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: Estrogen2018
Record Dates: First submitted 2018-10-22; First posted 2019-02-06 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Performance
Keywords: menstrual cycle; Estrogen; performance; variation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women using birth control
  Interventions: Other: estrogen level
- Women not using birthcontrol
  Interventions: Other: estrogen level

INTERVENTIONS:
Other: estrogen level — Women are tested at different times in their menstrual cycle, if there is a cohesion between performance and level of estrogen
  Other Names: Physical tests

SUMMARY:
This project aims to investigate if muscle strength and muscle power fluctuate during the menstrual cycle.

The hypothesis is that the greatest performance will be measured right before ovulation, and at it's lowest on day 1 and 2 of the menstrual cycle in women not using any form for hormonal protection.

And that the performance in women using birth control pills, not will variated in the period where they are taking pills (day 1-21).

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18-35 years of age
* BMI 18.5-25.

Exclusion Criteria:

* Smoking
* hormonal or metabolic disorders
* chronic sickness
* use of medication
* breast feeding, vegetarians
* diet containing a lot of soja based products
* injuries which make it impossible to do the tests

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women, 10 using 2. generations birth control pills and 30 not using any kind of hormonal protection.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in jumping height | 8 times per month, 2 to 5 days between measurements
  measuring of change in muscle power
Change in grip strength | 8 times per month, 2 to 5 days between measurements
  measuring of changes in muscle strength

SECONDARY OUTCOMES:
Change in hormone levels | 8 time per month, 2 to 5 days between measurements
  measuring of changes in hormone levels during cycle
Change in motivation by questionnaire | 8 times per month, 2 to 5 days between measurements
  measuring of changes in motivation for performing

CONTACTS AND LOCATIONS:
Locations (1):
- Section of Sport Science, Aarhus, Denmark

REFERENCES:
- [Derived] He W, Dam TV, Thogersen R, Hansen M, Bertram HC. Fluctuations in Metabolites and Bone Markers Across the Menstrual Cycle in Eumenorrheic Women and Oral Contraceptive Users. J Clin Endocrinol Metab. 2022 May 17;107(6):1577-1588. doi: 10.1210/clinem/dgac112. PMID 35213728